CLINICAL TRIAL: NCT03572387
Title: A Pilot Study of the Combination of 5-azacitidine (5-AZA) and All-trans Retinoic Acid (ATRA) for Prostate Cancer (PCa) With PSA-only Recurrence After Definitive Local Treatment
Brief Title: A Pilot Study of 5-AZA and ATRA for Prostate Cancer With PSA-only Recurrence After Local Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Vaibhav G Patel, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-0752
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Prostatic Neoplasms; Prostate Neoplasms; Prostate Cancer
Keywords: Prostate Neoplasms; Prostatic Neoplasms; 5-Azacitidine; all-trans retinoic acid; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Azacitidine; Tretinoin; Leuprolide

STUDY DESIGN:
Intervention Model Description: ll study enrollees will receive Lupron. After one month, they will be assigned in a 1:1 randomization to either the '5-AZA+ATRA' group or the 'delay therapy' group. Patients in the '5-AZA + ATRA' group will receive treatment on a 28-day cycle, in the absence of prohibitive toxicities, for 3 cycles. In the 'no therapy' group, patients will initially be observed for 3 cycles and then receive treatment for 3 cycles, in the absence of prohibitive toxicities. After the treatment period, all patients will be followed for up to 24 months from the start of the study or until the events leading to discontinuation are observed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5-AZA + ATRA ('early' 5-AZA+ATRA) (Experimental): Combination of 5-Azacitidine (5-AZA) + all trans retinoic acid (ATRA) group after one month of Lupron, group will receive treatment on a 28-day cycle, in the absence of prohibitive toxicities, for 3 cycles.
  Interventions: Drug: 5-Azacitidine; Drug: all trans retinoic acid; Drug: Lupron
- No therapy ('delayed' 5-AZA+ATRA) (Active Comparator): After one month of lupron, patients will receive no therapy for 3 cycles (12 weeks). After this observation period, patients will receive combination of 5-Azacitidine (5-AZA) + all trans retinoic acid (ATRA) group on a 28-day cycle, in the absence of prohibitive toxicities, for 3 cycles.
  Interventions: Drug: 5-Azacitidine; Drug: all trans retinoic acid; Drug: Lupron

INTERVENTIONS:
Drug: 5-Azacitidine — subcutaneously on days 1-5 at a dose of 40 mg/m^2
  Other Names: 5-AZA
Drug: all trans retinoic acid — 45 mg/m^2, will be taken orally on days 3-7 of each cycle, divided into two doses
  Other Names: ATRA
Drug: Lupron — 7.5 mg x 1
  Other Names: Leuprolide

SUMMARY:
This is a prospective, open-label, randomized, cross-over, pilot study of reprogramming therapy in patients with recurrent PCa based on rising PSA only. The primary objectives are to compare the disease progression-free rate at the end of 12 weeks of treatment between 5-AZA+ATRA and no therapy and to assess safety of the 5-AZA and ATRA combination. All study enrollees will receive Lupron. After one month, they will be assigned in a 1:1 randomization to either the '5-AZA+ATRA' group or the 'no therapy' group. Patients in the '5-AZA + ATRA' group will receive treatment on a 28-day cycle, in the absence of prohibitive toxicities, for 3 cycles. In the 'no therapy' group, patients will initially be observed for 3 cycles and then receive treatment for 3 cycles, in the absence of prohibitive toxicities. After the treatment period, all patients will be followed for up to 24 months from the start of the study or until the events leading to discontinuation are observed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Rising PSA
* PSADT ≤ 10 months prior to initiation of ADT
* No evidence of regional or active distant metastases, except for regional metastasis where salvage radiation therapy is not an option
* Indication for ADT after receiving definitive local therapy
* Males ≥ 18 years.
* ECOG performance status of ≤ 2
* Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy
* Ability to understand and the willingness to sign a written informed consent
* Ability to adhere to the study visit schedule and requirements of the protocol

Exclusion Criteria:

* Patients who have received ADT and/or other chemotherapy within 3 months prior to entering the study.
* Patients who have had radiotherapy or surgery within 4 weeks prior to entering the study. Minimally-invasive procedures for the purpose of diagnosis or staging of the disease are permitted.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-AZA and ATRA.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Significant active cardiac disease within the previous 6 months
* Inadequate organ and marrow function as defined below:
* leukocytes ≤ 3,000/mcL
* absolute neutrophil count ≤ 1,500/mcL
* platelets ≤ 100,000/mcl
* total bilirubin above normal institutional limits
* AST(SGOT)/ALT(SPGT) ≥ 2.5 X institutional upper limit of normal
* creatinine above normal institutional limits

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav G Patel, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected during the course of this clinical trial will primarily be shared with other investigators and health system staff, the IRB, FDA, and other reporting agencies, and/or transferred to other collaborators. Prior to transfer, the data collected must comply with, and must be limited by, the MSH's guidelines for Protecting the Rights and Privacy of Human Subjects.
Supporting Information: Study Protocol, ICF
Time Frame: 24 months
Access Criteria: At the end of study completion. It will be available for 5 years.

RESULTS

PARTICIPANT FLOW:
Groups:
- 'Early' 5-AZA+ATRA: Patients will receive Lupron 7.5 mg x 1. Four weeks later, they will receive 5-AZA+ATRA treatment on a 28-day cycle, in the absence of toxicities, for 3 cycles, followed by 3 cycles of observation
  Treatment:
  5-Azacitidine: subcutaneously on days 1-5 at a dose of 40 mg/m^2 all trans retinoic acid: 45 mg/m^2, will be taken orally on days 3-7 of each cycle, divided into two doses
- 'Delayed' 5-AZA+ATRA: Patients will receive Lupron 7.5 mg x 1. Four weeks later, they will undergo "observation" every 28 days for 3 cycles. Thereafter, patients will receive 5-AZA+ATRA treatment on a 28-day cycle, in the absence of toxicities, for 3 cycles.
  Treatment:
  5-Azacitidine: subcutaneously on days 1-5 at a dose of 40 mg/m^2 all trans retinoic acid: 45 mg/m^2, will be taken orally on days 3-7 of each cycle, divided into two doses
  -Taken for 3 cycles
Period: Treatment Phase 1 - 3 Cycles
Arm/Group | 'Early' 5-AZA+ATRA | 'Delayed' 5-AZA+ATRA
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0
Period: Treatment Phase 2 - 3 Cycles
Arm/Group | 'Early' 5-AZA+ATRA | 'Delayed' 5-AZA+ATRA
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 'Early' 5-AZA+ATRA: Patients will receive Lupron 7.5 mg x 1. Four weeks later, they will receive treatment on a 28-day cycle, in the absence of toxicities, for 3 cycles.
  Treatment:
  5-Azacitidine: subcutaneously on days 1-5 at a dose of 40 mg/m^2 all trans retinoic acid: 45 mg/m^2, will be taken orally on days 3-7 of each cycle, divided into two doses
  -Taken for 3 cycles
- Total: Total of all reporting groups
Arm/Group | 'Early' 5-AZA+ATRA | 'Delayed' 5-AZA+ATRA | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (6.8) | 71.8 (5.04) | 66.4 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 1 | 1 | 2
Gleason score [Count of Participants; unit: Participants] — grade of the cancer
  Participants
    <=7 (low to intermediate grade cancer) | 0 | 5 | 5
    >=8 (high grade cancer) | 5 | 3 | 8
    Unknown or Not Reported | 1 | 0 | 1
Prostate-Specific Antigen (PSA) doubling time [Mean (Standard Deviation); unit: months] | 3.51 (1.48) | 2.43 (1.06) | 2.89 (1.33)
PSA [Mean (Standard Deviation); unit: ng/ml] | 7.11 (11.7) | 2.99 (2.56) | 4.75 (7.81)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PSA Response
Description: Number of participants with PSA response, as defined by PSA decreased > 30% as compared from baseline.
Time Frame: baseline and 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 'Early' 5-AZA+ATRA | 'Delayed' 5-AZA+ATRA
Number analyzed (Participants) | 6 | 8
Participants | 0 | 0

2. Secondary Outcome: Percentage of Patients With Prolongation of PSA Doubling Time (PSADT) Post-treatment
Description: Percentage of patients with prolongation of PSA doubling time (PSADT) post-treatment compared to baseline after treatment with 3 cycles of Aza and ATRA.
Time Frame: baseline and 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 'Early' 5-AZA+ATRA | 'Delayed' 5-AZA+ATRA
Number analyzed (Participants) | 6 | 8
percentage of participants | 33.3 | 25

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | 'Early' 5-AZA+ATRA | 'Delayed' 5-AZA+ATRA
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 'Early' 5-AZA+ATRA (N=6) | 'Delayed' 5-AZA+ATRA (N=8)
Alanine Aminotransferrase increased (Investigations) | 2 | 0
Anemia (Investigations) | 4 | 3
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Aspartate Aminotransferase increased (Investigations) | 3 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Creatinine increased (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Edema Limbs (Vascular disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Generalized muscle weakness (General disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Headache (General disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Hot flashes (General disorders) | 2 | 2
Hypercalcemia (Investigations) | 1 | 0
Hyperglycemia (Investigations) | 5 | 3
Hyperkalemia (Investigations) | 0 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Cardiac disorders) | 2 | 0
Hypoalbuminemia (Investigations) | 1 | 0
Hyponatremia (Investigations) | 1 | 0
Immune system disorders other (Immune system disorders) | 0 | 1
Insomnia (General disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Pain (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Plaelet Count Decreased (Investigations) | 1 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1
Rectal pain (Gastrointestinal disorders) | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03572387/Prot_SAP_000.pdf